CLINICAL TRIAL: NCT06905106
Title: POlycythemia, Proteins and ErYthropoiesis
Acronym: POPEYE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GIRODON_2024
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Erythropoiesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with polycythemia: Whatever the origin of polycythemia
  Interventions: Biological: Collection of tube bottoms from blood samples taken in the clinic
- Patient controls: Patients with the same pathological features but without polycythemia
  Interventions: Biological: Collection of tube bottoms from blood samples taken in the clinic

INTERVENTIONS:
Biological: Collection of tube bottoms from blood samples taken in the clinic — Collection of tube bottoms from blood samples taken in the clinic

SUMMARY:
Erythropoiesis encompasses all the stages and mechanisms involved in the production of red blood cells, or erythrocytes, under the control of a large number of regulatory agents, most often proteins. Among these proteins, erythropoietin and interleukin-3 play a major role. Similarly, proteins involved in iron metabolism (erythroferrone, hepcidin, ferroportin, transferrin, ferritin) influence erythrocyte production more or less directly. The regulation of erythropoiesis is a fine, complex mechanism involving a large number of players, not only through the stimulation of hypoxia pathways to control erythropoietin synthesis, but also through the availability of iron, an essential element for erythropoiesis. Excessive erythrocyte production can lead to polycythemia, the causes of which are varied, primary or secondary, acquired or constitutional. The aim of this work is the descriptive study (quantitative and/or qualitative) of the various proteins involved in the regulation of erythropoiesis in patients with polycythemia. These proteins will be measured in the plasma of patients obtained after blood sampling or bloodletting (bloodletting being the most common treatment for polyglobulic patients) and will be compared with the proteins of patients without polycythemia.

ELIGIBILITY:
Inclusion Criteria:

- Persons who have given their non-opposition

Patients with polycythemia:

* haemoglobin value > 16 g/dl female or > 16.5 g/dl male
* with a well-identified cause: either primary (polycythemia Vaquez, erythropoietin receptor or LNK/SH2B3 mutation...) or secondary [cardio-respiratory pathologies, renal pathologies (post-transplant, polycystic kidney disease), metabolic pathologies, tumour (leiomyoma, pheochromocytoma...), constitutional mutations (hyperaffine haemoglobins, HIF2/EPAS1, PHD/EGLN1, VHL, ...)

Patients control:

- persons with a similar pathology to that of polycythemia patients, essentialy secondary, but without polycythemia, i.e. with a haemoglobin value of < 16 g/DL for women and < 16.5 g/DL for men

Exclusion Criteria:

* Person subject to a measure of legal protection (guardianship, tutorship)
* Person subject to a court order
* Pregnant, parturient or nursing woman
* Incapable of expressing consent
* Minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with polycythemia
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Measurement of various proteins involved in the regulation of erythropoiesis | at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France